CLINICAL TRIAL: NCT05279950
Title: Clinical and Patient Centred Outcome Performance of Full Mouth Ultrasonic Debridement Carried Out for the Treatment of Periodontitis Performed Either by Piezoelectric or Magnetostrictive Device. A Randomized Controlled Clinical Trial
Brief Title: Full Mouth Ultrasonic Debridement Carried Out Either by Piezoelectric or Magnetostrictive Device
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: University of Siena (Other)
Responsible Party: Principal Investigator, Nicola Discepoli, Professor, University of Siena
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: MAG001
Record Dates: First submitted 2020-03-04; First posted 2022-03-15 (Actual); Last update posted 2022-03-15 (Actual); Status verified 2022-03

CONDITIONS: Periodontitis, Adult
Keywords: periodontitis; patient centred outcomes; magnetostrictive
MeSH Terms: conditions — Chronic Periodontitis; Periodontitis | interventions — Emergency Treatment

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Piezoelectric (Active Comparator): Full-mouth ultrasonic debridement will be performed with a ultrasonic tip (vibration frequence >18 kHz) powered by a piezoelectric device
  Interventions: Device: Full-mouth ultrasonic debridement with piezoelectric device (EMS, mini piezon)
- Magnetostrictive (Experimental): Full-mouth ultrasonic debridement will be performed with a ultrasonic tip (vibration frequence >18 kHz) powered by a magnetostrictive device.
  Interventions: Device: Full-mouth ultrasonic debridement with magnetostrictive device (Cavitron Select, Dentsply)

INTERVENTIONS:
Device: Full-mouth ultrasonic debridement with piezoelectric device (EMS, mini piezon) — the use of ultrasonic oscillating tips allows supragingival and subgingival biofilm and dental calculus removal
  Arms: Piezoelectric
Device: Full-mouth ultrasonic debridement with magnetostrictive device (Cavitron Select, Dentsply) — the use of ultrasonic oscillating tips allows supragingival and subgingival biofilm and dental calculus removal
  Arms: Magnetostrictive

SUMMARY:
Treatment of periodontitis requires removal of dental biofilm both through professional mechanical plaque removal and domiciliar oral hygiene procedures. This study aims to compare biometric and psychological results after professional treatment of periodontitis carried out by piezoelectric or magnetostrictive ultrasonic devices.

DETAILED DESCRIPTION:
Patients diagnosed with periodontitis will be assessed for eligibility criteria. Full-mouth periodontal assessment will be performed by an examiner to detect severity and extension of the disease. Thereafter, patient will receive oral hygiene instruction and a closed envelope with patient allocation will be opened. After the allocation to the intervention group, full-mouth ultrasonic debridement will be delivered to the patient by an operator and information about patient perception will be collected. Three months later, patients will be recalled for a new periodontal assessment.

ELIGIBILITY:
Inclusion Criteria:

* >18 years
* periodontitis of stage 1 and 2
* absence of systemic chronic disease

Exclusion Criteria:

* anticoagulants treatment
* antibiotic treatment 3 months before the screening visit

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 52 (Estimated)
Dates: Start 2022-04-10 (Estimated); Primary Completion 2022-07-10 (Estimated); Study Completion 2022-10-30 (Estimated)

PRIMARY OUTCOMES:
Pain perception | through study completition, 1 year
  vas scale (0-10) for perception of pain after treatment
noise | through study completition, 1 year
  vas scale (0-10) for perception of noise after treatment
vibration | through study completition, 1 year
  vas scale (0-10) for perception of vibration after treatment

SECONDARY OUTCOMES:
pocket closure | through study completition, 1 year
  change of pocket probing depth (millimeter) after treatment measured with a periodontal probe

CONTACTS AND LOCATIONS:
Locations (1):
- AOUS, Siena, Italy

IPD SHARING:
Plan to Share IPD: No